CLINICAL TRIAL: NCT07073352
Title: Adverse Childhood Experiences and Premature Vascular Aging in Humans: The Role of SIRT1
Brief Title: ACEs, SIRT1, and Premature Vascular Aging in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nathaniel Jenkins (Other)
Responsible Party: Sponsor-Investigator, Nathaniel Jenkins, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 202407275
Record Dates: First submitted 2025-06-30; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Adverse Childhood Experiences; Endothelial Dysfunction
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicotinamide Riboside (Experimental): 4-weeks of twice daily, oral supplementation (2,000 mg/day) of NR (NIAGEN®
  , ChromaDEX, Irvine, CA).
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Placebo (Placebo Comparator): Participants randomized to the control group will consume matched placebo capsules containing microcrystalline cellulose.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Participants will consume 1,000 mg of nicotinamide riboside (NR) upon waking and with an evening meal, and complete a daily supplementation log to assist with compliance monitoring. NR is a naturally occurring vitamin B3 derivative readily taken up by cells as a direct NAD+ precursor. Similar NR supplementation protocols are well-tolerated, boost NAD+ concentrations by ~100-140% achieving a steady state within 1-2 weeks, and increase SIRT activity in humans.
  Arms: Nicotinamide Riboside
Dietary Supplement: Placebo — Participants will consume 1,000 mg of placebo (microcrystalline cellulose) upon waking and with an evening meal, and complete a daily supplementation log to assist with compliance monitoring.
  Arms: Placebo

SUMMARY:
Adverse childhood experiences (ACEs) are directly related to cardiovascular morbidity and mortality, and impaired vascular endothelial function (VEF) is an independent predictor of future cardiovascular disease (CVD) risk [1, 2]. Previous work from our lab (IRB 202010095) and others [3] demonstrates impaired VEF in young adults with prior exposure to ACEs even in the absence of clinical CVD risk factors. Sirtuin 1 (SIRT1) is a class III histone deacetylase (HDAC) that plays a role in regulating vascular homeostasis and reductions in SIRT1 are associated with age-related endothelial dysfunction [4]. We have shown that ACEs-related impairments in VEF are accompanied by reductions in SIRT1 [5]. However, the mechanisms by which ACE exposure promotes VEF remain unknown. The goal of this project is to establish proof of concept that alterations in vascular SIRT1 expression and activity mediate premature vascular aging in individuals with >=4 ACEs compared to those with 0 ACEs and that, because NAD+ is an essential substrate for SIRT1, increasing NAD+ bioavailability will restore VEF in those with >=4 ACEs.

Thus, we will use a robust translational approach coupling in vivo and in vitro measures of endothelial function, inflammation, oxidative stress, and SIRT1 expression and activity in young adults with (n=30-35) versus without (n=30-35) ACE exposure in a cross-sectional study, and during a randomized controlled trial employing a novel 4-week nicotinamide riboside (NR) supplementation approach to increase SIRT1 activity by increasing cellular NAD+ in ACE+ (n=15/group) to accomplish the following specific aims:

1. Determine the mechanisms by which ACE exposure alters the regulation of VEF by SIRT1. We hypothesize that compared to those without ACEs (ACE-), ACE+ will have (H1a) elevated endothelial oxidative stress and inflammation, (H1b) accompanied by reduced endothelial SIRT1 expression and increased p66SHC expression and acetylation of p65 and p53, (H1c) in association with lower VEF.
2. Determine how targeting SIRT1 by increasing NAD+ bioavailability affects VEF in young adults with ACEs. We hypothesize that systemic NR supplementation will (H2a) augment cellular SIRT1 activity and (H2b) improve VEF in ACE+.

[1] Felitti, V.J., Anda, R.F., Nordenberg, D., Williamson, D.F., Spitz, A.M., Edwards, V., Koss, M.P., & Marks, J.S. (1998). Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults: The adverse childhood experiences (ace) study. American Journal of Preventive Medicine, 14(4), 245-258. https://doi.org/10.1016/S0749-3797(98)00017-8. [2] Jenkins, N.D.M., & Robinson, A.T. (2022). How do adverse childhood experiences get under the skin to promote cardiovascular disease? A focus on vascular health. Function (Oxf), 3(4), zqac032. PMC9279110. 10.1093/function/zqac032. [3] Rodriguez-Miguelez, P., Looney, J., Blackburn, M., Thomas, J., Pollock, J.S., & Harris, R.A. (2022). The link between childhood adversity and cardiovascular disease risk: Role of cerebral and systemic vasculature. Function. 10.1093/function/zqac029. [4] Thompson, A. M., Wagner, R., & Rzucidlo, E. M. (2014). Age-related loss of SirT1 expression results in dysregulated human vascular smooth muscle cell function. American Journal of Physiology-Heart and Circulatory Physiology, 307(4), H533-H541. [5] Jenkins, N.D.M., Rogers, E.M., Banks, N.F., Tomko, P.M., Sciarrillo, C.M., Emerson, S.R., Taylor, A., & Teague, T.K. (2021). Childhood psychosocial stress is linked with impaired vascular endothelial function, lower sirt1, and oxidative stress in young adulthood. Am J Physiol Heart Circ Physiol, 321(3), H532-H541. PMC8461842. 10.1152/ajpheart.00123.2021

ELIGIBILITY:
Inclusion Criteria:

* 18 - 30 years
* ACE score of 0 OR ≥4 (Aim 1); ACE score ≥4 (Aim 2)

Exclusion Criteria:

* Resting arterial blood pressure >140/90 mmHg
* BMI ≥30 kg/m2 and/or weight unstable (>2.27 kg change) last 6 month
* Cardiovascular, metabolic, or pulmonary disease
* Cardiovascular or metabolic prescription drug use
* Vasoactive antidepressant drug use (SSRIs and clonidine)
* Currently pregnant or breastfeeding
* Heavy alcohol consumption (AUDIT screening)
* Use of illicit drugs
* Current tobacco use
* Regular vigorous (>6 MET s) aerobic exercise (>4 bouts/week, >30 min/bout)
* Dietary supplementation with antioxidants or habitual use of NSAIDs

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Vascular endothelial function | Before (0 Weeks) and after 4-week supplementation period (4 Weeks)
  Vascular endothelial function will be assayed in vivo using the brachial artery flow mediated dilation technique as the relative increase in brachial artery diameter in response to 5-minutes of forearm ischemia (peak - baseline diameter / baseline diameter * 100).

SECONDARY OUTCOMES:
Endothelial SIRT1 Expression | Before (0 Weeks) and after 4-week supplementation period (4 Weeks)
  Total SIRT1 Expression in Primary Endothelial Cells
Endothelial SIRT1 Activity | Before (0 Weeks) and after 4-week supplementation period (4 Weeks)
  Ratio of acetylated:total p53 in Primary Endothelial Cells
Cellular SIRT1 Activity in PBMCs | Before (0 Weeks) and after 4-week supplementation period (4 Weeks)
  Cellular SIRT1 activity from nuclear proteins in isolated peripheral blood mononuclear cells (ab156065).
Cellular NAD+ metabolites | Before (0 Weeks) and after 4-week supplementation period (4 Weeks)
  Semi-targeted high-resolution mass spectrometry will be used to quantify cellular levels of NAD+ and related metabolites, including: nicotinic acid adenine dinucleotide which is a highly sensitive marker of increased NAD+ metabolism via NR supplementation and adenosine diphosphate ribose which is an indicator of NAD+ consuming (SIRT) activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Laboratory of Applied Physiology and Lifestyle Medicine, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made publically available within 1 year of study completion. A study protocol paper will be published in 2026. The informed consent form will also be made publicly available at the award end date.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified data will be made publically available within 1 year of study completion in perpetuity.